CLINICAL TRIAL: NCT05762861
Title: Exploring Clinical Predictors of COPD Exacerbation in a Community Cohort
Acronym: EPISODE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Minho (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Maria Joao Barbosa, Principal investigator, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ISS 10805
Record Dates: First submitted 2021-06-20; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: COPD Exacerbation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual follow up (No Intervention): Group 1: To keep follow-up in their usual family practice/ pulmonology consultations
- Home telemonitoring (Experimental): Group 2: To keep follow-up in their usual family practice/ pulmonology consultations and associate an interactive home telemonitoring system managed by the researchers.
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Experimental — Patients will be every two weeks monitored by the researchers' team, taking into consideration lung function, symptoms, physical activity, pulse oximetry, body temperature, need for relief medication and Sputum characteristics. Over the 18 months, they will be the target of health education interventions, 2 individual and 2 in group.
  Other Names: Telemonitoring
  Arms: Home telemonitoring

SUMMARY:
The aim of our study is to assess the feasibility and benefits of the implementation of an interactive telemonitoring system for earlier detection of COPD exacerbations in a community cohort preventing further deterioration requiring hospital admissions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Aged 40 years or above
* Must be enrolled in health centres from Braga

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Number of COPD exacerbation with hospital admission | 18 months
Number of COPD exacerbation managed at home | 18 months
Quality of Life using St. George's Respiratory Questionnaire | 18 months
  Scores range from 0 (no effect on quality of life) to a maximum score of 100 (maximum perceived distress). A higher score means a poorer quality of life
Impact of COPD on patient's life using COPD Assessment Test (CAT) | 18 months
  Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Impact of the programme - rate of compliance | 18 months
  Measurement tool - questionnaire
Impact of the programme - satisfaction level | 18 months
  Measurement tool - questionnaire
Impact of the programme - % of retention of participating patients | 18 months
  Measurement tool - questionnaire

SECONDARY OUTCOMES:
Pulmonary function (FEV1 and FEV1/ FVC ratio after BD) | 18 months
Dyspnoea level (mMRC) | 18 months
Changes in GOLD classification | 18 months

IPD SHARING:
Plan to Share IPD: Undecided